CLINICAL TRIAL: NCT00843869
Title: Reversal of Tobacco-Related Sinusitis (Flight Attendant Medical Research Institute (FAMRI) Young Clinical Scientist Award)
Brief Title: Reversal of Tobacco-Related Sinusitis
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Flight Attendant Medical Research Institute (Other)
Responsible Party: Principal Investigator, Brad Woodworth, MD, Assistant Professor of Surgery, University of Alabama at Birmingham
Other Study IDs: F080623004
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Rhinosinusitis
MeSH Terms: conditions — Rhinosinusitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Zinc levels and hair samples will be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Rhinosinusitis: Participants with chronic rhinosinusitis

SUMMARY:
This study is focused on identifying the prevalence of passive or active smoke exposure and zinc deficiency in a cohort of patients who meet the objective and subjective guidelines for chronic rhinosinusitis set forth by the Sinus and Allergy Health Partnership.

DETAILED DESCRIPTION:
By using patient screening questionnaires and measuring hair nicotine, a well acknowledged biomarker of exposure to tobacco smoke, we will attempt a more objective study to examine the association between tobacco smoke and chronic rhinosinusitis. (CRS) Likewise, zinc deficiency is documented in numerous animal and human studies to decrease resistance to infectious diseases and is especially common among smokers. We will explore our hypothesis that SHS exposure and zinc deficiency contribute to CRS. To accomplish this, we will measure serum zinc and hair nicotine levels in CRS patients and correlate them to a variety of CRS diagnostic indicators. A second objective of this study is investigating alterations within the epithelium lining the sinonasal cavities in patients with chronic rhinosinusitis. The alterations may be one or a combination of anatomic, genetic, inflammatory, or infectious etiologies. To further investigate these possibilities we plan on taking residual clinical material from endoscopic sinus surgery specimens and performing various in vitro investigations including but not limited to microarray analysis, northern and western blot analysis, ciliary beat frequency analysis, immunohistochemistry, electron microscopy, and propagation of tissue with tissue culture techniques. Tissues taken from non-sinusitis patients undergoing sinonasal surgery will serve as a non-chronic rhinosinusitis control source of sinus mucosa.

ELIGIBILITY:
Inclusion Criteria:

* CRS and skull base surgery patients; CRS patients that meet the objective and subjective guidelines for CRS set forth by the Sinus and Allergy Health Partnership.

Exclusion Criteria:

* Ciliary dysfunction, autoimmune disease, CF or any known immunodeficiency.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic rhinosinusitis undergoing routine sinus and skull base surgery
Sampling Method: Non-Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2008-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
prevalence of passive or active smoke exposure | Completion of study
  This study is focused on identifying the prevalence of passive or active smoke exposure and zinc deficiency in a cohort of patients who meet the objective and subjective guidelines for chronic rhinosinusitis set forth by the Sinus and Allergy Health Partnership.

CONTACTS AND LOCATIONS:
Overall Officials: Brad Woodworth, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States